CLINICAL TRIAL: NCT06593639
Title: Does Prehabilitation be Able to Favorably Impact on the Pathway of Head and Neck Cancer Patients, Candidate to Surgery or Chemoradiotherapy as Primary Treatment? A Prospective Clinical Trial
Brief Title: Effect of Prehabilitation on Head and Neck Cancer Patients
Acronym: HNCANCERFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Deborah Locati (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Ospedaliero Universitaria di Sassari (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor-Investigator, Laura Deborah Locati, Head of Medical Oncology; Principal Investigator; Clinical Professor, Istituti Clinici Scientifici Maugeri SpA
Organization: Istituti Clinici Scientifici Maugeri SpA (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNRR-TR1-2023-12377022; PNRR-TR1-2023-12377022 (Other Grant/Funding Number: Italian Ministry of Health through PNRR resources (PNRR: M6/C2_CALL 2023))
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; prehabilitation; physical exercise; malnutrition; nutritional intervention; psychological support; cisplatin; hadrontherapy; ENT surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity; Malnutrition | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There will be two groups of head and neck cancer patients, one undergoing surgery plus (chemo)radiotherapy and the other undergoing definitive concomitant chemo-radiotherapy. Both groups will receive the prehabilitation intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery plus (chemo)radiotherapy (Experimental): Head and neck cancer patients undergoing surgery before (chemo)radiotherapy according to stage and risk factors.
  Interventions: Other: Prehabilitation before surgery
- Chemo-radiotherapy (Experimental): Head and neck cancer patients undergoing definitive concomitant chemo-radiotherapy (CRT) according to stage and risk factors.
  Interventions: Other: Prehabilitation before and during CRT

INTERVENTIONS:
Other: Prehabilitation before surgery — Prehabilitation multimodal program will start about 4 weeks before the surgery and will be continued until 2 weeks after the surgical intervention. Multimodal program comprises physical exercise, nutritional intervention, and psychological support provided before and during curative treatment for HNC patients.
  Other Names: physical exercise; nutritional intervention; psychological support
  Arms: Surgery plus (chemo)radiotherapy
Other: Prehabilitation before and during CRT — Prehabilitation multimodal program will start about 4 weeks CRT and will be continued in parallel until 2 weeks after the end. Multimodal program comprises physical exercise, nutritional intervention, and psychological support provided before and during curative treatment for HNC patients.
  Arms: Chemo-radiotherapy

SUMMARY:
The primary aim of the study is to investigate the feasibility of a prehabilitation program, which consists of a set of strategies including physical activity, nutritional support, and psychological counseling, carried out before and during cancer treatment for patients affected by head and neck tumors. About 4 weeks before surgery or the start of curative chemo-radiotherapy, the patient will begin the prehabilitation program, which will continue in parallel throughout the duration of the treatment and for up to 2 weeks after its completion. This prehabilitation program will include a combination of physical activity exercises, nutritional counseling, and psychological counseling sessions, all of which will be individualized for each patient. At the time of tumor diagnosis (T0), after 4 weeks of prehabilitation and before the start of the planned treatment (T1), 2 weeks after the end of treatment (T2), and after 6 months (T3), the patient will undergo a medical visit to collect anthropometric data, vital signs, a 6-minute walk test, and will complete a series of questionnaires aimed at assessing the risk of malnutrition, the development of anxiety and depression, and questionnaires to evaluate their quality of life. Throughout the duration of the study (i.e., up to T3, 6 months after the end of cancer treatment), the patient will wear an electronic watch, provided by the study, designed to measure vital signs, the number of daily steps, and the type and minutes of physical activity.

DETAILED DESCRIPTION:
Oncological prehabilitation is defined as the process within the care pathway that takes place between the moment of cancer diagnosis and the initiation of acute treatments. Prehabilitation aims to improve physical, emotional, and cognitive health before the start of cancer therapy, with the ultimate goal of preventing and reducing treatment-related comorbidities and mortality. It has also proven effective in reducing the adverse events of cancer therapies during the active phase of treatment, making it potentially useful at any stage of the care pathway for cancer patients. The role of exercise, nutrition, and stress reduction in improving outcomes for cancer patients has long been recognized in surgical prehabilitation, but the evidence for benefits in non-surgical cancer treatments is weaker due to fewer randomized clinical trials. Improvements in muscle strength, a reduction in cancer-related comorbidities (e.g., dyspnea, cardiotoxicity, urinary incontinence), and a positive impact on quality of life, including social well-being and a reduction in anxiety, depression, and stress, have been demonstrated. However, the literature regarding the role of multimodal prehabilitation in head and neck cancers is even weaker: there is limited data on feasibility and effectiveness, with most studies focusing on optimizing nutritional status in malnourished patients or improving dysphagia, but lacking data from prospective clinical trials. This study is designed as a prospective, multicenter, experimental, non-randomized, uncontrolled interventional trial. The objectives are: i) to evaluate the feasibility of prehabilitation before and during curative treatment for patients with head and neck cancer; ii) to investigate the efficacy outcomes of prehabilitation; iii) to conduct a cost-effectiveness analysis of prehabilitation.

Feasibility will be assessed by measuring patient acceptance, adherence, and satisfaction with the program. To evaluate adherence to the physical activity intervention, patients will be provided with wearable devices capable of measuring daily steps, type, and minutes of activity. To evaluate adherence to nutritional support, subjects will be asked to complete a food diary along with telephone interviews conducted by expert professionals. Adherence to psychological support requires a combination of self-reported measures, clinical evaluation, and behavioral observation. A patient will be considered adherent if they complete at least 80% of the assigned tasks. The investigators will consider prehabilitation feasible if more than 50% of patients in the treatment group adhere to the program for the entire scheduled period. To investigate the efficacy of the treatment, validated questionnaires on quality of life and the patient's health status will be administered. Secondary endpoints will include the difference between questionnaire scores at the end versus the beginning of the intervention in terms of variables quantifying the response to cancer treatments and the patient's physiological status. It will also be possible to calculate both the cost-effectiveness and cost-utility balance of the intervention, considering the difference between the intervention arm and the historical control arm in terms of quality-adjusted life years. The activities carried out to achieve this objective will allow us to characterize the changes between the start and end of the intervention. Any significant (positive or negative) variation between the start and end of the intervention will be considered a result.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Candidate to curative treatment (platinum-based chemoradiotherapy or surgery + RT +/- CT)
* ECOG PS 0-1
* Fit for prehabilitation program (medical, physical, and mental conditions that don't contraindicate physical exercise and oral nutrition)
* Ability to understand and adhere to exercise or lifestyle modifications
* Date of treatment beginning no later than 60 days from baseline assessment
* Provide valid informed consent prior to any study procedure

Exclusion Criteria:

* Unstable medical condition requiring immediate attention (e.g uncontrolled heart failure; unstable angina; severe respiratory distress) must prioritize
* Patients with very advanced stage of disease, candidate to palliative treatment
* Uncontrolled cancer symptoms or pain
* Need for early treatment initiation
* Frailty subjects: patients with severe functional impairment
* Significant muscle wasting, limiting the participation in prehabilitation exercise
* Severe cognitive or mental health issues, precluding prehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of multimodal prehabilitation | From enrollment to the end of prehabilitation program, 2 weeks after the end of curative treatment
  The feasibility will be measured by the rate of adherence to prehabilitation interventions. To assess the adherence to the physical activity intervention, the investigators will equip patients with commercially available activity trackers. Patients will wear the activity tracker until 6 months after the end of treatment. To assess the adherence to the nutritional intervention a telephone 24-hour dietary recall (24HR) interview will be employed. 24HR is a retrospective method that monitors and assesses the food and drinks consumption of the subjects during the previous day. Adherence to psycho-oncological support requires a combination of self-report measure, clinical assessment and behavioral observation. The three reports will be aggregated to a one reported value: a patient will be considered adherent to prehabilitation program if they will be adherent to each intervention.
Efficacy of multimodal prehabilitation | From enrollment to 2 weeks after the end of oncological treatment
  A comparison between T0 (cancer diagnosis) and the other time points (T1: after 4 weeks of prehabilitation, T2: 2 weeks after the end of oncological treatments, T3: at 6 months of follow-up) will be made to exploit any differences. To test the efficacy of physical activity, the functional capacity over time will be monitored, measuring as the difference in absolute change in 6-minute walk distance (6MWD) between T0 and T1 and between T0 and T2. In addition, the Handgrip strength (HGS) will be employed as a biomarker of overall health status. Two questionaries (i.e. NRS-2002 and MUST) will be used as screening tools to exploit the risk of malnourishment. ASonA, Distress Thermometer, and FACT- HN will be used to test the psycho-oncological intervention efficacy. The three reports will be aggregated to a one reported value: the program will be considered effective if each intervention will be effective.
Cost-effectiveness of multimodal prehabilitation | From the enrollment to 6 months after the end of the oncological treatment
  To evaluate the sustainability, the cost-utility analysis of the prehabilitation intervention will be evaluated. Cost Utility Analysis is an economic analysis comparing the incremental cost of a program to the incremental health improvement in terms of quality adjusted life years (QALYs). The EORTC QLQ-C30 questionnaire will be used to predict EQ-5D-5L through a mapping algorithm, which is one of the most used instrument for measuring QALYs.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Istituto Nazionale Tumori IRCCS, Fondazione G. Pascale, Napoli, Italy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
  - Istituti Clinici Scientifici Maugeri, Pavia, Italy
  - National Center of Adrotherapy Oncology, Pavia, Italy
  - Azienda Ospedaliero Universitaria di Sassari, Sassari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cantwell LA, Fahy E, Walters ER, Patterson JM. Nutritional prehabilitation in head and neck cancer: a systematic review. Support Care Cancer. 2022 Nov;30(11):8831-8843. doi: 10.1007/s00520-022-07239-4. Epub 2022 Aug 1. PMID 35913625
- [Background] Loughney L, West MA, Moyses H, Bates A, Kemp GJ, Hawkins L, Varkonyi-Sepp J, Burke S, Barben CP, Calverley PM, Cox T, Palmer DH, Mythen MG, Grocott MPW, Jack S; Fit4Surgery group. The effects of neoadjuvant chemoradiotherapy and an in-hospital exercise training programme on physical fitness and quality of life in locally advanced rectal cancer patients: a randomised controlled trial (The EMPOWER Trial). Perioper Med (Lond). 2021 Jun 22;10(1):23. doi: 10.1186/s13741-021-00190-8. PMID 34154675
- [Background] Urvaylioglu AE, Kutluturkan S, Kilic D. Effect of Kegel exercises on the prevention of urinary and fecal incontinence in patients with prostate cancer undergoing radiotherapy. Eur J Oncol Nurs. 2021 Apr;51:101913. doi: 10.1016/j.ejon.2021.101913. Epub 2021 Feb 15. PMID 33639454
- [Background] Halkett G, O'Connor M, Jefford M, Aranda S, Merchant S, Spry N, Kane R, Shaw T, Youens D, Moorin R, Schofield P; RT Prepare project team. RT Prepare: a radiation therapist-delivered intervention reduces psychological distress in women with breast cancer referred for radiotherapy. Br J Cancer. 2018 Jun;118(12):1549-1558. doi: 10.1038/s41416-018-0112-z. Epub 2018 Jun 1. PMID 29855611
- [Background] Goldsmith I, Chesterfield-Thomas G, Toghill H. Pre-treatment optimization with pulmonary rehabilitation in lung cancer: Making the inoperable patients operable. EClinicalMedicine. 2020 Nov 30;31:100663. doi: 10.1016/j.eclinm.2020.100663. eCollection 2021 Jan. PMID 33554075
- [Background] Quist M, Langer SW, Lillelund C, Winther L, Laursen JH, Christensen KB, Rorth M, Adamsen L. Effects of an exercise intervention for patients with advanced inoperable lung cancer undergoing chemotherapy: A randomized clinical trial. Lung Cancer. 2020 Jul;145:76-82. doi: 10.1016/j.lungcan.2020.05.003. Epub 2020 May 8. PMID 32416432
- [Background] Lippi L, Turco A, Moalli S, Gallo M, Curci C, Maconi A, de Sire A, Invernizzi M. Role of Prehabilitation and Rehabilitation on Functional Recovery and Quality of Life in Thyroid Cancer Patients: A Comprehensive Review. Cancers (Basel). 2023 Sep 10;15(18):4502. doi: 10.3390/cancers15184502. PMID 37760472
- [Background] Howe L, Husband A, Robinson-Barella A. Prescribing pre- and post-operative physical activity interventions for people undergoing breast cancer surgery: A qualitative systematic review. Cancer Med. 2024 Feb;13(4):e7063. doi: 10.1002/cam4.7063. PMID 38457236
- [Background] Voorn MJJ, Driessen EJM, Reinders RJEF, van Kampen-van den Boogaart VEM, Bongers BC, Janssen-Heijnen MLG. Effects of exercise prehabilitation and/or rehabilitation on health-related quality of life and fatigue in patients with non-small cell lung cancer undergoing surgery: A systematic review. Eur J Surg Oncol. 2023 Oct;49(10):106909. doi: 10.1016/j.ejso.2023.04.008. Epub 2023 May 2. PMID 37301638
- [Background] Waterland JL, McCourt O, Edbrooke L, Granger CL, Ismail H, Riedel B, Denehy L. Efficacy of Prehabilitation Including Exercise on Postoperative Outcomes Following Abdominal Cancer Surgery: A Systematic Review and Meta-Analysis. Front Surg. 2021 Mar 19;8:628848. doi: 10.3389/fsurg.2021.628848. eCollection 2021. PMID 33816546
- [Background] Sabajo CR, Ten Cate DWG, Heijmans MHM, Koot CTG, van Leeuwen LVL, Slooter GD. Prehabilitation in colorectal cancer surgery improves outcome and reduces hospital costs. Eur J Surg Oncol. 2024 Jan;50(1):107302. doi: 10.1016/j.ejso.2023.107302. Epub 2023 Nov 28. PMID 38043359
- [Background] Molenaar CJL, Minnella EM, Coca-Martinez M, Ten Cate DWG, Regis M, Awasthi R, Martinez-Palli G, Lopez-Baamonde M, Sebio-Garcia R, Feo CV, van Rooijen SJ, Schreinemakers JMJ, Bojesen RD, Gogenur I, van den Heuvel ER, Carli F, Slooter GD; PREHAB Study Group. Effect of Multimodal Prehabilitation on Reducing Postoperative Complications and Enhancing Functional Capacity Following Colorectal Cancer Surgery: The PREHAB Randomized Clinical Trial. JAMA Surg. 2023 Jun 1;158(6):572-581. doi: 10.1001/jamasurg.2023.0198. PMID 36988937
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Silver JK, Flores LE. Integrating Prehabilitation into the Cancer Survivorship Framework. Eur Urol Focus. 2024 Jan;10(1):23-25. doi: 10.1016/j.euf.2023.11.006. Epub 2023 Nov 22. PMID 37996272
- [Background] Carli F, Silver JK, Feldman LS, McKee A, Gilman S, Gillis C, Scheede-Bergdahl C, Gamsa A, Stout N, Hirsch B. Surgical Prehabilitation in Patients with Cancer: State-of-the-Science and Recommendations for Future Research from a Panel of Subject Matter Experts. Phys Med Rehabil Clin N Am. 2017 Feb;28(1):49-64. doi: 10.1016/j.pmr.2016.09.002. PMID 27913000
- [Background] Ligibel JA, Bohlke K, May AM, Clinton SK, Demark-Wahnefried W, Gilchrist SC, Irwin ML, Late M, Mansfield S, Marshall TF, Meyerhardt JA, Thomson CA, Wood WA, Alfano CM. Exercise, Diet, and Weight Management During Cancer Treatment: ASCO Guideline. J Clin Oncol. 2022 Aug 1;40(22):2491-2507. doi: 10.1200/JCO.22.00687. Epub 2022 May 16. PMID 35576506
- [Background] Silver JK, Baima J. Cancer prehabilitation: an opportunity to decrease treatment-related morbidity, increase cancer treatment options, and improve physical and psychological health outcomes. Am J Phys Med Rehabil. 2013 Aug;92(8):715-27. doi: 10.1097/PHM.0b013e31829b4afe. PMID 23756434